CLINICAL TRIAL: NCT06244030
Title: The Effect of Core Stabilization Exercises on Trunk Muscle Strength, Upper Extremity Performance and Spinal Stability in Female Wrestlers
Brief Title: The Effect of Core Stabilization Exercises in Female Wrestlers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Emine Atıcı, Principal Investigator, Okan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 011
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Exercise Addiction; Trunk Muscle Strength; Upper Extremity; Wrestling

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core Stabilization Group (Experimental): The athletes in the core stabilization group will be applied a 15-20 repetition core stabilization exercise program 3 days a week for 6 weeks by the researcher. The duration of the exercise program is planned not to exceed 30 minutes. The values before and after the exercise program will be recorded.
  Interventions: Other: core stabilization group
- Control Group (No Intervention): The control group will not be given any exercise other than their own wrestling training program.

INTERVENTIONS:
Other: core stabilization group — The athletes in the training group will be applied 15-20 repetitions of core stabilization exercise program 3 days a week for 6 weeks by the researcher.
  Arms: Core Stabilization Group

SUMMARY:
This study was planned to investigate the effect of core stabilization exercise program on trunk muscle strength, spinal stability and upper extremity performance in elite wrestling athletes.

ELIGIBILITY:
Inclusion Criteria:

* Being between 14 and 21 years old and interested in wrestling
* Actively pursuing a life of wrestling
* Participate in training at least 4 days a week
* Wrestling in freestyle style.
* To confirm that there is no injury problem
* Being a licensed athlete

Exclusion Criteria:

* Experiencing any serious injury problems

Ages: 14 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Assessment of muscle strength | ''6 weeks''
  An isokinetic dynamometer will be used for trunk muscle strength assessment.
Medicine Ball Throwing Test | ''6 weeks''
  This test is used to determine limb strength and power. The materials needed will be a 2.5 kg medicine ball and a meter. The individual will be asked to stand one step behind the starting line with the medicine ball in participant hand. When the ball is at chest level, the individual will be asked to take a step and throw the ball as far as participant can. Scoring will be done by measuring the distance the ball falls from the starting line
Closed Kinetic Chain Upper Limb Test | ''6 weeks''
  This test will measure upper extremity strength, endurance and closed kinetic chain stability. Two athletic bands and a stopwatch will be needed for this test measurement. Two pieces of athletic tape will be placed on the floor at 0.9 meter intervals. The person will be asked to take a push-up position with participant hands open at the level of the band. The person will be asked to move his/her hands from one band line to the other as fast as possible and touch each line by moving like a "wiper". The touches will be counted for 15 seconds with a stopwatch. Power scores will be determined by taking 68% of the person's body weight (the weight of the upper extremities, head and trunk at the upper level) in kilograms and multiplying it by the number of touches and dividing the result by 15.
Upper extremity Y balance test | ''6 weeks''
  Functional dynamic postural balance assessments of individuals will be performed with the Y balance test. Scores on the Y balance test kit are based on three directions will be recorded. The Y balance Test kit will be used in medial, superolateral and inferolateral directions with 120° angles between them. With the hand tested on the test kit in the push-up position with the tested hand in the center of the device at the junction of the angles, the participants will be asked to take the Y balance test box to the fingertip of the other hand to the farthest point they can reach and return it to its original position, and the distance they can reach will be measured in cm. Measurements will be taken bilaterally with three repetitions. After obtaining the mean values, normative values will be obtained by dividing the sum of right and left by two

SECONDARY OUTCOMES:
Functional Reach Test | ''6 weeks''
  In this test researchers will ask participant to stand sideways next to a wall and make a fist with the arm close to the wall and keep it parallel to the floor. researchers will mark the 3rd metacarpal head on the wall. Meanwhile, researchers will ask the person to reach forward as far as they can without taking a step and mark the new 3rd metacarpal head. Researchers will measure the distance between the marked lines at the beginning and end. Researchers will make 3 attempts and finish the test by averaging the last 2 attempts

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Okan University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Will be shared when necessary